CLINICAL TRIAL: NCT01702623
Title: A Single Dose, Two-Period, Two-Treatment, Two-Sequence Crossover Bioequivalence Study of Oxcarbazepine 600 mg Suspension Under Fasted Conditions
Brief Title: Crossover Bioequivalence Study of Oxcarbazepine 600 mg Suspension Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OXCA-S600-PVFS-2
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures | interventions — Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxcarbazepine first, then Trileptal (Active Comparator): Single dose of oxcarbazepine suspension, 600 mg, then single dose of trileptal suspension, 600 mg (after washout period)
  Interventions: Drug: Oxcarbazepine
- Trileptal first, then Oxcarbazepine (Active Comparator): Single dose of oxcarbazepine suspension, 600 mg, then single dose of trileptal suspension, 600 mg (after washout period
  Interventions: Drug: Oxcarbazepine

INTERVENTIONS:
Drug: Oxcarbazepine
  Other Names: Trileptal

SUMMARY:
The objective of this study was to prove the bioequivalence of Roxane Laboratories' Oxcarbazepine Suspension 600 mg under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to oxcarbazepine or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 10 Days

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Zamora, MD, Principal Investigator — Worldwide Clinical Trials Drug Development Solutions (formerly CEDRA Clinical Research)
Locations (1):
- Worldwide Clinical Trials Drug Development Solutions (formerly CEDRA Clinical Research), San Antonio, Texas, United States